CLINICAL TRIAL: NCT00179816
Title: High-Dose Chemotherapy With Tandem Peripheral Blood Stem Cell (PBSC) Rescue for the Treatment of High-Risk Pediatric Solid Tumors.
Brief Title: Tandem Peripheral Blood Stem Cell (PBSC) Rescue for High Risk Solid Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Morris Kletzel, Children's Memorial Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMT 0499 Solid
Record Dates: First submitted 2005-09-10; First posted 2005-09-16 (Estimated); Last update posted 2010-10-11 (Estimated); Status verified 2010-10

CONDITIONS: Ewing's Sarcoma; Soft Tissue Sarcoma; Hepatoblastoma; Hodgkin's Disease; Germ Cell Tumor
Keywords: wilm's tumor; stem cell transplantation; solid tumor
MeSH Terms: conditions — Sarcoma, Ewing; Sarcoma; Hepatoblastoma; Hodgkin Disease; Neoplasms, Germ Cell and Embryonal; Wilms Tumor | interventions — Drug Therapy; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: High-Dose Chemotherapy with Tandem PBSC Rescue. — Patients on this study will undergo a tandem Peripheral Blood Stem Cell Rescue following high-dose chemotherapy. The first Peripheral Blood Stem Cell Rescue will consist of Etoposide, Carboplatin, Cyclophosphamide, and Mesna. Once the patient recovers, the patient will be evaluated again and will then undergo a second stem cell transplant consisting of the chemotherapy drugs; Melphalan, Cyclophosphamide, and Mesna.
  Other Names: Cyclophosphamide call also be referred to as Cytoxan

SUMMARY:
This study uses a double autologous peripheral blood stem cell rescue (PBSC) following dose-intensive chemotherapy for the treatment of high-risk pediatric solid tumors.

DETAILED DESCRIPTION:
Significant advances have been made in recent years in the treatment of solid tumors of childhood. However, much of the improvement in survival has been made in low stage and localized disease. Of significance is the fact that the improvements have come in up-front remission rates without translation into significantly high event-free survival(EFS) or overall survival (OS). This is despite the fact that these tumors as a whole are largely chemotherapy responsive.

Recent advances in the understanding of the biology of hematopoeitic stem cells have driven the design of treatment regimens that allow for dose intensification without unacceptable hematologic toxicity. Protocol development has focused on active agents that have a broad range between hematologic and non-hematologic toxicities. This study uses a double autologous peripheral blood stem cell rescue (PBSC) following dose-intensive chemotherapy for the treatment of high-risk pediatric solid tumors. This study utilizes PBSC to limit the risk of tumor cell contamination while retaining prompt hematologic recovery from these highly intensified treatments.

ELIGIBILITY:
Inclusion Criteria:

* Malignant Diseases:

  * Ewing's sarcoma/PNET:

    * CR1 - Metastatic disease at diagnosis, tumor volume > 100 ml, pelvic bone primary
    * CR2 - Locally recurrent disease
  * Soft tissue sarcoma

    * CR1 - Metastatic disease at diagnosis or locally advanced disease where local control is suboptimal (i.e., inability to provide radiation therapy due to extent of disease).
    * CR2 - Locally recurrent disease (VGPR2 acceptable)
  * Hepatoblastoma:

    * VGPR1 - Patients with metastatic disease at diagnosis who have a persistently elevated alpha FP, or unresectable primary as a way of converting to resectable.
    * CR2/VGPR2
  * Hodgkin's Disease:

    * VGPR1 - Progression on primary therapy/Refractory disease
    * CR2/VGPR2
  * Germ Cell Tumor:

    * CR2/VGPR2 - recurrent disease
  * Wilms Tumor:

    * CR2/VGPR2 - recurrent disease
* IRB approved signed written informed consent by patient and/or their legally authorized guardian.
* Patients 21 years of age or younger at initial diagnosis, with older patients considered individually for primary pediatric disease diagnosis.
* Adequate central venous access (double lumen CVL or 2 single lumen PCVC).
* Adequate PBSC harvests with a minimum of 2.0 x 108 MNC/kg available for each PBSC rescue.
* Organ Function:

  * Platelets > 50,000/ml
  * SGOT < 10 x upper limits of normal
  * Creatinine < 1.5 x normal baseline
  * Normal cardiac function in accordance with institutional policies
  * Normal pulmonary function in accordance with institutional policies.
* Physiologic status:

  * No active infections
  * Adequate performance status as measured by Karnofsky (> 70%) or Lansky scale (> 60%) as appropriate for age.
* Bone Marrow Status

  * No evidence of morphologic involvement with tumor at the time of transplant

Off Study Criteria:

* Severe toxicity. Contact the Study Coordinator immediately and complete Adverse Reaction Form.
* Disease progression or relapse prior to PBSC #1 or between PBSC rescue # 1 and #2.
* Inability to collect adequate numbers of PBSC for successful transplantation.
* Patient or parent/guardian refusal to remain on study.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Estimated)
Dates: Start 1999-04; Primary Completion 2012-09 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Determine the feasibility and toxicity of tandem PBSC rescue following high dose chemotherapy as consolidation in pediatric patients with high risk solid tumors. | annually

SECONDARY OUTCOMES:
Evaluate length of remission and long term disease free survival in chemotherapy responsive high-risk pediatric solid tumor patients treated using this approach. | Annually
Evaluate correlation between cell dose and time to engraftment in high-risk pediatric solid tumor patients treated using this approach. | Time to engraftment

CONTACTS AND LOCATIONS:
Overall Officials: Morris Kletzel, M.D., Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Children's Memorial Hospital, Chicago, Illinois, United States